CLINICAL TRIAL: NCT03296592
Title: Predictive Value of Diffusion MRI in Cervical Spondylotic Myelopathy
Brief Title: Diffusion MRI in Cervical Spondylotic Myelopathy (CSM)
Acronym: CSM
Status: Active, not recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Wilson Z. Ray, Principal Investigator, Washington University School of Medicine
Other Study IDs: NS047592-10-201706177
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cervical Spondylotic Myelopathy
Keywords: myelopathy; diffusion MRI; spinal cord injury; spinal cord compression; spondylosis; cervical
MeSH Terms: conditions — Spinal Cord Diseases; Spinal Cord Injuries; Spinal Cord Compression; Spondylosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Investigational subjects: Patients who have been diagnosed with cervical spondylotic myelopathy and who will be undergoing surgical correction for this diagnosis.
  Visit 1 Investigational subjects will undergo a clinical assessment. Patients will undergo a DBSI MRI
  Visit 2. 6 months after surgery, investigational subjects will undergo a clinical assessment.
  Visit 3 12 months after surgery, investigational subjects will undergo a clinical assessment
  Visit 4 18 months after surgery, investigational subjects will undergo a clinical assessment.
  Visit 5 24 months after surgery, investigational subjects will undergo a clinical assessment and a DBSI MRI.
  Interventions: Diagnostic Test: MRI with DBSI technology
- Control group: Healthy volunteers aged 45-65 Visit 1: DBSI MRI Visit 2: 24 months after first MRI, patient will undergo the second MRI
  Interventions: Diagnostic Test: MRI with DBSI technology

INTERVENTIONS:
Diagnostic Test: MRI with DBSI technology — The MRI will be done with diffusion basis spectrum imaging

SUMMARY:
Patients who have been diagnosed with Cervical Spondylotic Myelopathy will be asked to undergo an MRI using diffusion basis spectrum imaging (DBSI) technology. The patients will have this MRI preoperatively and at 24 months postop. The investigators believe that with this imaging, biomarkers will be able to be seen to assist in prediction of long term outcomes in patients with spinal cord compression. These patients will be compared to healthy cohorts who will also undergo an MRI using the DBSI technology.

DETAILED DESCRIPTION:
CSM is the most common form of spinal cord injury and is the leading cause of progressive disability in patients over the age of 65. A major shortcoming limiting the clinical management of CSM is the lack of quantifiable metrics to 1) base clinical decisions and 2) predict potential for functional recovery following surgical intervention. DBSI MRI will provide imaging biomarkers to more reliably predict a patient's clinical course, response to therapy, and long-term prognosis.

Patients who are diagnosed with CSM will have an MRI using the DBSI technology preoperatively and at 24 months. Surgical patients will be assessed with the Neck Disability Index (NDI), Disability of the Arm, Shoulder and Hand (DASH), hand grip dynamometer and Manual Muscle Testing (MMT), the modified Japanese Orthopaedic Association scale (mJOA), and the Major Depression Inventory (MDI), the Short Form-36 (SF-36) and Nurick scoring.

A control group of healthy volunteers will have an MRI using the DBSI technology when enrolled and then again between 12-24 months later.

ELIGIBILITY:
Inclusion Criteria:

* History of ongoing spinal cord compression,
* clinical evidence of CSM as determined by signs and symptoms including, but not limited to loss of manual dexterity, extremity weakness, sensory abnormalities, quadriparesis, loss of proprioception, and positive Babinski's or Hoffman's sign.

Exclusion Criteria:

* pregnant
* having an MRI incompatible device
* having a known diagnosis of amyotrophic lateral sclerosis, multiple sclerosis, rheumatoid arthritis, concomitant thoracic and/or lumbar stenosis, spine tumor or HIV-related myelopathy and having systemic instability or being deemed unable to tolerate standard MRI sequencing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enroll from our patient population and 20 patients from healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Accurate prediction of neurologic outcomes after surgery | 24 months
  Outcome measure will assess spinal cord DBSI pathological metrics at baseline and at 24 months.

SECONDARY OUTCOMES:
Assessment of effects of blood flow deficits on spinal cord pathology | 24 months
  Outcome measure will assess effects of blood flow deficits on spinal cord pathology and determine the accuracy of axonal loss quantification in CSM

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Z Ray, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
The investigators will not share individual participant data with other researchers. Aggregate data will be made available at study completion.